CLINICAL TRIAL: NCT01079312
Title: Patient-controlled Sedation vs Propofol Infusion for ERCP:a Randomized Controlled Study
Brief Title: Patient-controlled Sedation With Propofol and Remifentanyl for Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maxim Mazanikov, M.D., Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: a001c; 2008-007968-42 (EudraCT Number)
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography
Keywords: ERCP; patient-controlled sedation; propofol; remifentanil; sedation level
MeSH Terms: interventions — Infusion Pumps; Propofol; Fentanyl; Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol infusion (Active Comparator): Anaesthesiologist's managed intravenous infusion of propofol 10mg/ml
  Interventions: Device: infusion pump; Drug: propofol; Drug: fentanyl
- Patient-controlled sedation (Active Comparator): self-administration of propofol and remifentanil mixture during ERCP
  Interventions: Device: infusion pump for patient-controlled sedation; Drug: propofol; Drug: sedative mixture; Drug: remifentanil hydrochlorid

INTERVENTIONS:
Device: infusion pump — anaesthesiologist´s managed infusion of propofol 10 mg/ml at rate of 10-60ml/h during ERCP targeting to moderate sedation level
  Other Names: -Braun AG; -an infusion pump
  Arms: Propofol infusion
Device: infusion pump for patient-controlled sedation — self-administration of propofol and remifentanil mixture with zero lockout time and without dose limit and background infusion via Arcomed,Syramed AG,Switzerland self-administration pump.
  Other Names: -Arcomed,Syramed AG,Switzerland; -infusion pump designed for self administration of the drugs
  Arms: Patient-controlled sedation
Drug: propofol — Propofol 10 mg/ml solution is a short-acting, intravenously administered hypnotic agent.In propofol infusion group moderate sedation was initiated with propofol 40 mg bolus,thereafter propofol infusion was started at rate of 0.5 mg/kg/h.If the performance of ERCP become difficult infusion rate was increased gradually ad maximum rate of 9 mg/kg/h.Additional propofol boluses of 20-40 mg were available in both groups due to an anaesthesiollogist´s ´desigion.In patient-controlled sedation group propofol was used for preparation of sedative mixture.
  Other Names: -Diprivan; -Recofol; -Fresofol
Drug: fentanyl — Fentanyl citrate 50 mcg/ml,solution for injection,is a narcotic analgesic.In propofol infusion group 0.05 mg of fentanyl was administered intravenously before initiation of sedation. Additional 0.05 mg boluses of fentanyl were given if nociceptive stimulus was anticipated.
  Other Names: -fentanyl citrate; -fentanyl
  Arms: Propofol infusion
Drug: sedative mixture — Sedative mixture was prepared by adding 5 ml of remifentanil hydrochlorid solution (50 mcg/ml)to 20 ml of propofol (10 mg/ml)
  Other Names: -Ultiva; -Diprivan
  Arms: Patient-controlled sedation
Drug: remifentanil hydrochlorid — Solution of remifentanil hydrochlorid (50 mcg/ml) was used for preparation of sedative mixture(see sedative mixture for details)
  Other Names: -Ultiva
  Arms: Patient-controlled sedation

SUMMARY:
Background: Deep sedation with propofol and opioid is commonly used for endoscopic retrograde cholangiopancreatography (ERCP), but is associated with increased morbidity and mortality. Delivery of propofol and short-acting potent opioid analgesic using a self-administration device (patient-controlled sedation, PCS) could be another option for this purpose. Comparative studies with PCS for ERCP are lacking.The main objective of this prospective randomized trial trial was to compare PCS with propofol/remifentanil to anaesthesiologist managed propofol sedation during ERCP.

DETAILED DESCRIPTION:
80 elective ERCP patients were randomized to anaesthesiologist managed propofol sedation (PI-group) or PCS with propofol/remifentanil (PCS-group). Sedation degree was estimated every 5 min throughout the procedure using Ramsay´s and Gillham´s sedation scores. Total amount of propofol was calculated at the end of procedure. Endoscopists´ and patients´ satisfaction was evaluated with questionary.

ELIGIBILITY:
Inclusion Criteria:

* elective ERCP-patients

Exclusion Criteria:

* allergy to propofol or opioid;
* ASA-class (American Society of Anaesthesiology) greater than 3;
* inability to co-operate;
* drugs abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
propofol and opioid consumption | one day
  total consumption of propofol,milligramms and opioid,microgramms during ERCP procedure
vital signs | one day
  heart rate,blood pressure,peripheral oxygen saturatuion,breathing rate,expiratory carbon dioxide concentration
patient´s and endoscopist´s satisfaction | one day
  Likert scale 1-7

SECONDARY OUTCOMES:
sedation level | one day
  sedation level assested with Ramsay,Gillham,OAA/S sedation scores

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Mazanikov, MD, Principal Investigator — Helsinki University Central Hospital,Department of Anaesthesiology; Marianne Udd, MD, PhD, Principal Investigator — Helsinki University Central Hospital,Department of Surgery; Outi Lindström, MD, Principal Investigator — Helsinki University Central Hospital,Department of Surgery; Leena Kylänpää, Docent, Principal Investigator — Helsinki University Central Hospital,Department of Surgery; Pekka Aho, MD, PhD, Principal Investigator — Helsinki University Central Hospital,Department of Vascular Surgery; Jorma Halttunen, Docent, Principal Investigator — Helsinki University Central Hospital,Department of Surgery; Martti Färkilä, Professor, Principal Investigator — Helsinki University Central Hospital,Department of Gasroenterology; Reino Pöyhiä, Docent, Study Chair — Helsinki University Central Hospital,Department of Anaesthesiology
Locations (1):
- Helsinki University Central Hospital,Meilahti hospital,Endoscopy unit, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No
Due to Finnish legal restriction patient data can not be accessed by others but the researches

REFERENCES:
- [Result] Mazanikov M, Udd M, Kylanpaa L, Lindstrom O, Aho P, Halttunen J, Farkkila M, Poyhia R. Patient-controlled sedation with propofol and remifentanil for ERCP: a randomized, controlled study. Gastrointest Endosc. 2011 Feb;73(2):260-6. doi: 10.1016/j.gie.2010.10.005. PMID 21295639